CLINICAL TRIAL: NCT04470037
Title: Multidisciplinary Study of Novel NMDA Modulation for Neurodegenerative Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Hsien-Yuan Lane, Director, Department of psychiatry, China Medical University Hospital, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH105-REC1-023
Record Dates: First submitted 2020-05-26; First posted 2020-07-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease With Dementia
Keywords: Parkinson's disease; Dementia; NMDA; DAAOI
MeSH Terms: conditions — Parkinson Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAAOI-P (Experimental): DAAOI-P 250-1500mg
  Interventions: Drug: DAAOI-P
- Starch pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DAAOI-P — DAAOI-P 250-1500mg
  Arms: DAAOI-P
Drug: Placebo — starch pill
  Arms: Starch pill

SUMMARY:
Alzheimer's disease (AD) and Parkinson's disease (PD) are currently the leading neurodegenerative disorders. Considering the fact that aged population is rapidly growing, it has become a critical issue to find more effective medications for these two disorders. The aim of this project is to examine the effectiveness and safety of DAAOI-P treatment for PD with dementia.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) and Parkinson's disease (PD) are currently the leading neurodegenerative disorders. Despite some therapeutic benefits from the medications targeting at cholinergic and dopaminergic pathways in AD and PD respectively, it remains far away from a satisfied treatment goal. DAAOI-P is a D-amino acid oxidase (DAAO) inhibitor and an agent specific to facilitate NMDA receptor subunit 1 (NR1). The investigators have demonstrated that NMDA-enhancement can help PD-D patients. The aim of this project is to examine the effectiveness and safety of DAAOI-P treatment for PD with dementia. In addition to evaluating clinical treatment response, multidisciplinary examinations, including electroencephalography, transcranial magnetic stimulation, magnetic resonance imaging (MRI), and psychophysical methods to analyze the changes in perceptual sensitivity to faces, emotion expressions, and biological motion recognition will be arranged to elucidate the underlying mechanism of NMDA modulation in neurodegenerative disorder.

ELIGIBILITY:
Inclusion Criteria:

* PD-D will be diagnosed according to the criteria proposed by Movement Disorder Society task force statement. (Emre et al. 2007) . The following wordings are modified from the task force statement. I. Core features

  1. Diagnosis of PD according to Queen Square Brain Bank criteria
  2. A dementia syndrome with insidious onset and slow progression, developing within the context of established PD and diagnosed by history, clinical, and mental examination, defined as:

     * Impairment in more than one cognitive domain
     * Representing a decline from premorbid level
     * Deficits severe enough to impair daily life, independent of the impairment ascribable to motor or autonomic symptoms
     * MMSE score between 10-26.

II. Associated clinical features

1. Cognitive features: Impaired attention, executive functions, visuo-spatial functions or memory. Core functions of language are largely preserved.
2. Behavioral features:

   * Apathy
   * Changes in personality and mood
   * Hallucination• Delusions
   * Excessive daytime sleepiness

III. Features which do not exclude PD-D, but make the diagnosis uncertain

* Co-existence of any other abnormality which may by itself cause cognitive impairment, but judged not to be the cause of dementia.
* Time interval between the development of motor and cognitive symptoms is uncertain

IV. Features suggesting other conditions or diseases as cause of mental impairment, which, when present make it impossible to reliably diagnose PD-D

* Cognitive and behavioral symptoms appearing solely in the context of other conditions such as:

  1. Acute confusion due to systemic illnesses or drug intoxication.
  2. Major depression
* Features compatible with "Probable Vascular dementia" criteria according to NINDS-AIREN Criteria for the diagnosis of probable and possible PD-D [Probable PD-D] Both core features must be present. In associated clinical features, typical profile of cognitive deficits should be present in at least 2 of the 4 core cognitive domains. The presence of at least one behavioral symptom supports the diagnosis of probable PD-D. None of group III and IV features is present. [Possible PD-D] Both core features must be present. In associated clinical features, the cognitive impairment is atypical in one or more domains. The behavioral symptoms are not necessary to be present. One or more of the group III features may be present. No group IV feature is allowed to be present.

Exclusion Criteria:

1. Patients with uncontrollable malignancy, severe heart failure, uremia under hemodialysis, or decompensated liver cirrhosis.
2. Patients taking anticholinergics within 30 days of recruitment.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
The improvement of gait and neuropsychiatric symptoms | week 0, 8, 16, 24
  Change in Unified Parkinson's Disease Rating Scale (UPDRS)
  UPDRS: Unified Parkinson's Disease Rating Scale Minimum value: 0 Maximum value: 199 The higher score means a worse outcome.

SECONDARY OUTCOMES:
Gait function | week 0, 8, 16, 24
  The Cyclogram of Gait
  Minimum value: 0 Maximum value: 100 The higher score means a better outcome.
Fall assessment | week 0, 8, 16, 24
  The fall assessment test of China Medical University Hospital
  Minimum value: 0 Maximum value: 10 The higher score means a worse outcome.
Cognitive function | week 0, 8, 16, 24
  Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog)
  ADAS-Cog: Alzheimer's Disease Assessment Scale-Cognitive Subscale Minimum value: 0 Maximum value: 70 The higher score means a worse outcome.
Neuropsychiatric symptoms | week 0, 8, 16, 24
  Change in Neuropsychiatry Inventory (NPI)
  NPI: Neuropsychiatry Inventory Minimum value: 0 Maximum value: 144 The higher score means a worse outcome
The improvement of Parkinson's disease | week 0, 8, 16, 24
  Change in The 39-item Parkinson's Disease Questionnaire (PDQ-39)
  PDQ-39: The 39-item Parkinson's Disease Questionnaire Minimum value: 0 Maximum value: 156 The higher score means a worse outcome.
Behavioral Pathology of dementia | week 0, 8, 16, 24
  Change in Behavioral Pathology in Alzheimer's Disease Rating Scale (Behave-AD)
  Behave-AD: Behavioral Pathology in Alzheimer's Disease Rating Scale Minimum value: 0 Maximum value: 75 The higher score means a worse outcome.
Severity of dementia | week 0, 8, 16, 24
  Change in Clinical Dementia Rating (CDR)
  CDR: Clinical Dementia Rating Minimum value: 0 Maximum value: 5 The higher score means a worse outcome.
Neuroimaging examinations | week 0, 24
  Neuroimaging examinations contains: (1) Structural MRI, (2) Resting-state fMRI, and (3) Working memory fMRI.
Face perception | week 0, 8, 16, 24
  Changes in perceptual discriminability (d-prime index)
  Minimum value: 0 (chance level); Maximum value: 3.0 (nearly perfect)
Emotion recognition and imitation | week 0, 8, 16, 24
  Changes in emotion recognition accuracy and imitation probability
  Minimum value: 0%; Maximum value: 100% (Higher score indicate a better outcome)
Transcranial magnetic stimulation | week 0, 8, 16, 24
  Change in Transcranial Magnetic Stimulation (TMS) assessments
Electroencephalography | week 0, 8, 16, 24
  Changes in Mismatch negativity (MMN)

CONTACTS AND LOCATIONS:
Overall Officials: Lane, Principal Investigator — Department of Psychiatry, China Medical University Hospital
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan